CLINICAL TRIAL: NCT01545661
Title: A Randomised Control Trial of Sputum Induction, and New and Emerging Technologies in a High HIV Prevalence Primary Care Setting
Brief Title: Utility of Sputum Induction and Novel Technologies to Improve TB Diagnosis in a High HIV Prevalence Primary Care Setting
Acronym: SINET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Jonathan Peter, Dr, University of Cape Town
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: SINET study
Record Dates: First submitted 2011-07-07; First posted 2012-03-07 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; diagnosis; sputum induction; primary care
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sputum induction (Experimental): Enrolled patients receive sputum induction (using ultrasonic nebulisation with hypertonic saline)
  Interventions: Procedure: Sputum induction
- No sputum induction (Active Comparator): Enrolled patients randomised to this study arm will receive an observed expectorated sputum collection attempt. Research nurses train study patients on the method of producing sputum spontaneously.
  Interventions: Procedure: standard routine expectorated sputum

INTERVENTIONS:
Procedure: Sputum induction — Ultrasonic nebulisation 3% hypertonic saline nebulised for duration of 20 mins
  Arms: Sputum induction
Procedure: standard routine expectorated sputum — Patients in the control group are trained by the research staff to produce sputum but no device is utilized. Sputum is spontaneously expectorated where possible
  Arms: No sputum induction

SUMMARY:
This study will investigate the benefit of using Sputum induction for TB diagnosis in a primary care clinic for adult TB suspects that are either unable to produce a sputum sample (sputum scarce) or on initial diagnostic work-up have 2 negative sputum smear samples (WHO standard for frontline TB diagnosis). The investigators hypothesize that acquiring an induced sputum sample for smear microscopy and liquid TB culture will decrease time-to-diagnosis and time-to-treatment initiation in smear negative/sputum scarce TB patients in a primary care clinic in a resource-limited high TB HIV prevalent setting.

DETAILED DESCRIPTION:
Tuberculosis is on the increase in Africa. A key area of weakness in TB control efforts is the inability to make a rapid diagnosis. This is, in part, due to the inability to obtain representative biological samples and the non-availability of cheap, effective, rapid and field-friendly diagnostic tools. Indeed, in HIV positive patients, where the sensitivity of sputum smear is as low as 20%, culture results take several weeks and a significant proportion of patients do not expectorate sputum. Sputum induction for the diagnosis of TB has been evaluated in several studies, has been shown to have a good yield, feasibility and safety when performed correctly, and with diagnostic comparability to bronchoscopy. Few studies have evaluated the performance of induced sputum outside of the hospital environment and the tolerability, yield and performance outcome of sputum induction in a primary care facility has yet to be evaluated. The objective of this study is two-fold. We seek to evaluate, through a randomized controlled trial, the feasibility, performance outcomes and impact on time-to-diagnosis and -treatment of sputum induction, in a high HIV prevalence primary care setting, for the diagnosis of smear negative/ sputum scarce TB. We hypothesize that acquiring an induced sputum sample for smear microscopy and liquid TB culture will decrease time-to-diagnosis and time-to-treatment initiation in smear negative/sputum scarce TB patients in a primary care clinic in a resource-limited high TB HIV prevalent setting. We will also evaluate the potential incremental benefit of novel technologies to improve the rapidity and diagnostic yield using induced sputum samples (Xpert MTB/RIF assay, microscopic observation drug susceptibility testing (MODS) and the Genotype MTB DRplus line probe assay).

ELIGIBILITY:
Inclusion Criteria:

1. 2x smear negative or sputum scarce TB suspects
2. Primary care patient (not referred by doctor)
3. Adult patients (>18 years)
4. Able to provide informed consent

Exclusion Criteria:

1. Not meeting inclusion criteria
2. <18 years
3. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2009-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Time-to-treatment initiation | Up to 48 days after enrollment
  Time-specific proportion of patients initiated on TB treatment between study arms Time-points to be analysed include 3, 5, 7, 10, 14, 21, 48 days from enrollment.

SECONDARY OUTCOMES:
Diagnostic yield of sputum culture | Up to 2 months after enrollment
  Difference in diagnostic yield of a single sputum TB culture between study arms.
  This will compare the single induced or expectorated sputum sample collected at study enrollment.
Diagnostic yield and accuracy of sputum smear microscopy | Up to 2 months after enrollment
  Difference in diagnostic yield and accuracy of a single sputum TB smear between study arms.
  This will compare the single induced or expectorated sputum sample collected at study enrollment.
  Liquid TB culture will be used as the reference standard for assessment of diagnostic accuracy Fluorescence smear microscopy will be performed on auramine-O stained concentrated samples
Feasibility of sputum induction in primary care clinics | 2 years
  Feasibility and robustness of performing sputum induction in primary care clinics (measures include - sputum induction failure rates, turn-around-time, user appraisals and evaluation)
Safety and tolerability of sputum induction performed in primary care clinics | 2 years
  Side-effects of sputum induction procedures Number of induced sputum procedures terminated because of patient side-effects and safety
Diagnostic yield and accuracy of additional diagnostics including Xpert MTB/RIF assay, MODS and Genotype MTBDRplus | 2 years
  Difference in diagnostic yield and accuracy of Xpert MTB/RIF, MODS liquid culture and the Genotype MTBDRplus on a single induced or expectorated sputum sample collected at enrollment.
  Liquid TB culture will be used as the reference standard for diagnostic accuracy measures.
Cost-analysis of sputum induction for primary care clinics | 2 years
  Based on diagnostic accuracy measures of different diagnostic tests between the induced sputum and standard care groups, cost-of-diagnosis will be calculated and compared

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan G Peter, MBChB, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Peter JG, Theron G, Pooran A, Thomas J, Pascoe M, Dheda K. Comparison of two methods for acquisition of sputum samples for diagnosis of suspected tuberculosis in smear-negative or sputum-scarce people: a randomised controlled trial. Lancet Respir Med. 2013 Aug;1(6):471-8. doi: 10.1016/S2213-2600(13)70120-6. Epub 2013 Jul 19. PMID 24429245